CLINICAL TRIAL: NCT02855749
Title: Comparison of 3 Techniques for Percutaneous Tracheostomy : Traditional Marking Technique, Ultrasonography Guided Long Axis Approach and Short Axis Approach
Brief Title: Ultrasound Guided Percutaneous Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERZINCAN UNIVERSITY 2
Record Dates: First submitted 2016-07-31; First posted 2016-08-04 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Reliability of the Ultrasound in Percutaneous Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- landmark group (No Intervention): percutaneous tracheostomy with traditional landmark technique
- ultrasound-guided long axis group (Active Comparator): percutaneous tracheostomy will be implemented In the real-time ultrasound-guided in plane technique
  Interventions: Procedure: ultrasound-guided percutaneous tracheostomy
- ultrasound-guided short axis group (Active Comparator): percutaneous tracheostomy will be implemented In the real-time ultrasound-guided out of plane technique
  Interventions: Procedure: ultrasound-guided percutaneous tracheostomy

INTERVENTIONS:
Procedure: ultrasound-guided percutaneous tracheostomy — to compare the reliability of the traditional landmark method, ultrasound-guided long axis in plane applications and ultrasound-guided short-axis out of plane application in the implementation process percutaneous tracheostomy
  Arms: ultrasound-guided long axis group; ultrasound-guided short axis group

SUMMARY:
Use of the ultrasound before, during and after percutaneous tracheostomy allows us great advantages; anatomy of the pre and paratracheal region and displaying potential aberrant vessels, and so the needle and dilator to move away from risk areas and ensure the prevention of possible vascular complications. Measuring the distance from the skin into the trachea can be done and this allows us to choose the average size tracheostomy tube.

The aim of this study, In the process of applying percutaneous tracheostomy, to compare the reliability of the traditional landmark method, ultrasound-guided long axis in plane application and ultrasound-guided short axis out of plane application.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients in intensive care
* the decision to open percutaneous tracheostomy
* over 18 years

Exclusion Criteria:

* under 18 years
* Patients with high or unstable intracranial pressure
* Patients with severe coagulation disorders
* Patients attached collar
* hemodynamically unstable patients, despite the use of high doses of vasoactive drugs
* patients with infections in tracheostomy area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The success of the first application | ten minute
successful tube placement rate | fifteen minüte
Complications during the procedure | one month

SECONDARY OUTCOMES:
The number of puncture | ten minute
total tracheostomy application time | fifteen minute
Early and late complications after the process | one month

CONTACTS AND LOCATIONS:
Overall Officials: İlke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Delaney A, Bagshaw SM, Nalos M. Percutaneous dilatational tracheostomy versus surgical tracheostomy in critically ill patients: a systematic review and meta-analysis. Crit Care. 2006;10(2):R55. doi: 10.1186/cc4887. PMID 16606435
- [Result] Cheung NH, Napolitano LM. Tracheostomy: epidemiology, indications, timing, technique, and outcomes. Respir Care. 2014 Jun;59(6):895-915; discussion 916-9. doi: 10.4187/respcare.02971. PMID 24891198
- [Result] Simon M, Metschke M, Braune SA, Puschel K, Kluge S. Death after percutaneous dilatational tracheostomy: a systematic review and analysis of risk factors. Crit Care. 2013 Oct 29;17(5):R258. doi: 10.1186/cc13085. PMID 24168826
- [Result] McCormick B, Manara AR. Mortality from percutaneous dilatational tracheostomy. A report of three cases. Anaesthesia. 2005 May;60(5):490-5. doi: 10.1111/j.1365-2044.2005.04137.x. PMID 15819770
- [Result] Flint AC, Midde R, Rao VA, Lasman TE, Ho PT. Bedside ultrasound screening for pretracheal vascular structures may minimize the risks of percutaneous dilatational tracheostomy. Neurocrit Care. 2009 Dec;11(3):372-6. doi: 10.1007/s12028-009-9259-z. Epub 2009 Aug 13. PMID 19680824
- [Result] Rudas M. The role of ultrasound in percutaneous dilatational tracheostomy. Australas J Ultrasound Med. 2012 Nov;15(4):143-148. doi: 10.1002/j.2205-0140.2012.tb00197.x. Epub 2015 Dec 31. PMID 28191160
- [Result] Chacko J, Nikahat J, Gagan B, Umesh K, Ramanathan M. Real-time ultrasound-guided percutaneous dilatational tracheostomy. Intensive Care Med. 2012 May;38(5):920-1. doi: 10.1007/s00134-012-2514-3. Epub 2012 Feb 17. No abstract available. PMID 22349428
- [Result] Rajajee V, Fletcher JJ, Rochlen LR, Jacobs TL. Real-time ultrasound-guided percutaneous dilatational tracheostomy: a feasibility study. Crit Care. 2011;15(1):R67. doi: 10.1186/cc10047. Epub 2011 Feb 22. PMID 21342494
- [Derived] Kupeli I, Nalbant RA. Comparison of 3 techniques in percutaneous tracheostomy: Traditional landmark technique; ultrasonography-guided long-axis approach; and short-axis approach - Randomised controlled study. Anaesth Crit Care Pain Med. 2018 Dec;37(6):533-538. doi: 10.1016/j.accpm.2017.11.011. Epub 2017 Dec 7. PMID 29225012